CLINICAL TRIAL: NCT03534713
Title: Phase III Study Comparing Neoadjuvant Chemotherapy With Carboplatin and Paclitaxel Followed by Standard Therapy, With Standard Therapy Alone in Women With Cervical Cancer and Para Aortic Positive Lymph Node.
Brief Title: Induction Chemotherapy Followed by Standard Therapy in Cervical Cancer With Aortic Lymph Node Spread
Acronym: ONCOCOL01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/17/0213
Record Dates: First submitted 2018-04-16; First posted 2018-05-23 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cervical Cancer TNM Staging Regional Lymph Nodes (N)
Keywords: Neoadjuvant chemotherapy; Cervical Cancer; Paraaortic Lymph Node Involvement; Carboplatin; Paclitaxel
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Carboplatin; Paclitaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant chemotherapy+standard therapy (Experimental): neoadjuvant chemotherapy with carboplatin aera Under curve 5 and paclitaxel 175 mg/m² every 21 days during 3 cycles followed by standard therapy with extended field external radiotherapy and concomitant chemotherapy (Cisplatin 40mg/m2 weekly)
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Cisplatin; Radiation: Radiotherapy
- standard therapy alone (Active Comparator): standard therapy with extended field external radiotherapy and concomitant chemotherapy (Cisplatin 40mg/m2 weekly)
  Interventions: Drug: Cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Carboplatin — carboplatin aera Under curve 5 on day 1, every 21 days during 3 cycles
  Other Names: Carbo
  Arms: Neoadjuvant chemotherapy+standard therapy
Drug: Paclitaxel — paclitaxel 175 mg/m² on day 1, every 21 days during 3 cycles
  Other Names: Taxol
  Arms: Neoadjuvant chemotherapy+standard therapy
Drug: Cisplatin — Cisplatin 40mg/m² given once a week during 5 weeks
  Other Names: Platinol
Radiation: Radiotherapy — 45 gray to the pelvis and para aortic area over 5 weeks + intracavitary brachytherapy alone or prior to surgery, depending on response to treatment according to the current guidelines
  Other Names: radiation therapy

SUMMARY:
The main objective of this study is to determine whether neoadjuvant chemotherapy with Carboplatin and paclitaxel plus standard cisplatin-based chemoradiation with extended fields improves overall survival rates compared to standard therapy alone in women with cervical cancer with paraaortic lymph node involvement.

Women in the experimental arm will receive neoadjuvant chemotherapy with carboplatin and paclitaxel every 21 days during 3 cycles followed by standard therapy with extended field external radiation therapy and concomitant chemotherapy. Women in the control arm will receive standard therapy with extended field external radiation therapy and concomitant chemotherapy.

310 patients will be recruited during 4.5 years, with 3 years of follow up period.

DETAILED DESCRIPTION:
The survival outcome of patients with carcinoma of the cervix and positive paraaortic lymph node is poor and the potential benefit of neoadjuvant chemotherapy before extended field chemoradiotherapy has never been assessed.

Paraaortic nodal spread in cervical cancer is a blind spot in the management of cervical cancer. It is necessary to evaluate additional treatment.

While the presence of paraaortic nodal metastases often indicates occult systemic disease, the investigators continue to treat them as a loco-regional disease.

Using neoadjuvant chemotherapy, improvement of overall survival rates is expected in women with cervical cancer and para-aortic positive lymphadenopathy without increasing the incidence of further toxicity.

The propose is to determine whether neoadjuvant chemotherapy with Carboplatin and paclitaxel plus standard cisplatin-based chemoradiation with extended fields improves overall survival rates compared to standard therapy alone in women with cervical cancer with paraaortic lymph node involvement.

Secondary objectives will be to compare progression free survival, acute and long term toxicities, patterns of disease recurrence and patient quality of life between arms This is a phase III, multicenter, randomized, open label study, recruiting 310 patients during 4.5 years, with 3 years of follow up period.

Two groups will be compared : neoadjuvant chemotherapy with Carboplatin and paclitaxel plus standard cisplatin-based chemoradiation with extended fields, versus standard therapy alone.

Randomization will be stratified according to International federation of gynecology and obstetrics stages at diagnosis (IB1, IB2, IIA versus IIB-IVA), the size of positive para aortic lymphadenopathy and the number of node involved and will be balanced by blocks.

Women in the experimental arm will receive neoadjuvant chemotherapy with carboplatin and paclitaxel followed by standard therapy with extended field external radiation therapy and concomitant chemotherapy then intracavitary brachytherapy, alone or prior to surgery, depending on response to treatment according to the current guidelines.

Women in the control arm will receive standard therapy with extended field external radiation therapy and concomitant chemotherapy then brachytherapy, alone or prior to surgery, depending on response to treatment according to the current guidelines.

Follow up will be the same between arms. But in experimental arm, during treatment phase, a clinical examination and biological assessment will be performed before each cycle of neoadjuvant chemotherapy. Therefore, at the end of neoadjuvant treatment, just before standard treatment magnetic resonance imaging and positron emission tomography-computed tomography will be performed.

Then, all Participants will be followed every 4 months until 2 years after randomization and every 6 months during the third year according to current follow-up guideline for cervical cancer. Disease response and disease progression will be assessed using clinical examination. Quality of life will be estimated at baseline, at the end of neoadjuvant chemotherapy, before intracavitary brachytherapy and at each follow-up visit until 3 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically proven invasive carcinoma of the uterine cervix and para aortic lymphadenopathy determined by either a positive positron emission tomography with 2-deoxy-2-[fluorine-18]fluoro- D-glucose integrated with computed tomography or if negative positron emission tomography computed tomography based on histological examination of paraaortic lymph node dissection.
* Performance status Eastern Cooperative Oncology Group 0-2
* Stage International Federation of Gynecology and Obstetrics IB1 to IVA at diagnosis with para-aortic lymph node involvement
* Adenocarcinoma or squamous cell carcinoma or adenosquamous carcinoma
* Adequate renal function (creatinine clearance ≥60 mL/min)
* Adequate hepatic function (bilirubin <1.5 times normal and Serum Glutamooxaloacetate Transferase < 3 times normal)
* Adequate hematopoietic function Platelet count > 100x10 9/l and Absolute neutrophil count > 1.5X10 9/l)
* Written Informed consent for participation

Exclusion Criteria:

* Stage Federation of Gynecology and Obstetrics IVB at diagnosis
* Others histologies than adenocarcinoma, squamous cell carcinoma and adenosquamous carcinoma.
* Women who receive any prior chemotherapy for her cervical cancer
* Pregnant or lactating women
* Prior ( within the last 5 years) malignancies other than non-melanoma skin cancer
* Inadequate renal, hepatic or hematopoietic function (Cf previously)
* Cardiovascular pathology New York Heart Association II or more
* Pre-existing Peripheral neuropathy Common toxicity Criteria grade ≥ 2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3 years
  time between random assignment and death resulting from any cause

SECONDARY OUTCOMES:
progression free survival | fron date of randomization until the date of first documented progression or date of death from any cause, assessed up to 3 years
  time from randomization to first documentation of disease progression or death due to any cause.
adverse events | 3 years
  classified using the Common Terminology Criteria for Adverse Events and coded using Medical Dictionary for Regulatory Activities dictionary Pattern of disease recurrence will include locoregional recurrence and distant metastasis
quality of life questionnaire C30 and CX24 | 3 years
  assessed using the European Organization for Research and Treatment Quality of Life Questionnaire C30 and CX24, all subscales responses will be converted to 0 to 100 scales according to European Organization for Research and Treatment guidelines
patterns of first relapse | 3 years
  location of relapse or metastasis by magnetic resonance imaging

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie MOTTON, MD, Principal Investigator — University Hospital, Toulouse
Locations (11):
- France (11):
  - CHU de Bordeaux, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - CHI Créteil, Créteil
  - Institut Paoli Calmettes, Marseille
  - CH Lyon Sud, Pierre-Bénite
  - CHU de Poitiers, Poitiers
  - Institut de Cancérologie de l'Ouest - Nantes, Saint-Herblain
  - CHU La Réunion, Saint-Pierre
  - Clinique Pasteur, Toulouse
  - University Hospital Toulouse, Toulouse
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grigsby PW, Heydon K, Mutch DG, Kim RY, Eifel P. Long-term follow-up of RTOG 92-10: cervical cancer with positive para-aortic lymph nodes. Int J Radiat Oncol Biol Phys. 2001 Nov 15;51(4):982-7. doi: 10.1016/s0360-3016(01)01723-0. PMID 11704321
- [Background] Varia MA, Bundy BN, Deppe G, Mannel R, Averette HE, Rose PG, Connelly P. Cervical carcinoma metastatic to para-aortic nodes: extended field radiation therapy with concomitant 5-fluorouracil and cisplatin chemotherapy: a Gynecologic Oncology Group study. Int J Radiat Oncol Biol Phys. 1998 Dec 1;42(5):1015-23. doi: 10.1016/s0360-3016(98)00267-3. PMID 9869224
- [Background] Chantalat E, Vidal F, Leguevaque P, Lepage B, Mathevet P, Deslandres M, Motton S. Cervical cancer with paraaortic involvement: do patients truly benefit from tailored chemoradiation therapy? A retrospective study on 8 French centers. Eur J Obstet Gynecol Reprod Biol. 2015 Oct;193:118-22. doi: 10.1016/j.ejogrb.2015.07.017. Epub 2015 Aug 5. PMID 26295788
- [Background] Duenas-Gonzalez A, Zarba JJ, Patel F, Alcedo JC, Beslija S, Casanova L, Pattaranutaporn P, Hameed S, Blair JM, Barraclough H, Orlando M. Phase III, open-label, randomized study comparing concurrent gemcitabine plus cisplatin and radiation followed by adjuvant gemcitabine and cisplatin versus concurrent cisplatin and radiation in patients with stage IIB to IVA carcinoma of the cervix. J Clin Oncol. 2011 May 1;29(13):1678-85. doi: 10.1200/JCO.2009.25.9663. Epub 2011 Mar 28. PMID 21444871
- [Background] Singh RB, Chander S, Mohanti BK, Pathy S, Kumar S, Bhatla N, Thulkar S, Vishnubhatla S, Kumar L. Neoadjuvant chemotherapy with weekly paclitaxel and carboplatin followed by chemoradiation in locally advanced cervical carcinoma: a pilot study. Gynecol Oncol. 2013 Apr;129(1):124-8. doi: 10.1016/j.ygyno.2013.01.011. Epub 2013 Jan 24. PMID 23353129